CLINICAL TRIAL: NCT04520542
Title: The Effect of Acupressure Application on Menopausal Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adiyaman University Research Hospital (Other)
Responsible Party: Principal Investigator, Didem Kucukkelepce, Lokman Hekim University, Adiyaman University Research Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Supportive Care
Other Study IDs: Lokman Hekim Universty
Record Dates: First submitted 2020-08-16; First posted 2020-08-20 (Actual); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: Menopausal Syndrome

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- acupressure (Experimental): The application was performed on the determined acupressure points by considering the direction of the meridian in a certain order. It was performed with the administration order of Spleen 6th point (SP 6) and Large Intestine 4th point (Li 4). In total, the administration was performed with 4 acupressure points including 2 points in the upper/lower extremity along with the parallel points in each intervention. Each acupressure point was massaged for 30 seconds to provide circulation before the pressure. After the massage, consecutive pressures were applied for 90 seconds. In each intervention, a total of 8-minute sessions were applied to 4 points as 2 minutes for each point. Consecutive pressures were applied on a frequency that did not disturb the women, did not cause pain, and had a soothing effect. Until the end of the intervention it was continued 2 times a week, 16 times in total in 8 weeks.
  Interventions: Other: Acupressure Application
- Control Group (No Intervention): no intervation

INTERVENTIONS:
Other: Acupressure Application — Acupressure was administered in a semi-sitting or supine position where the woman felt comfortable and the researcher could perform the practice comfortably to the acupressure points. The application was performed on the determined acupressure points by considering the direction of the meridian in a certain order. It was performed with the administration order of Spleen 6th point (SP 6) and Large Intestine 4th point (Li 4). In total, the administration was performed with 4 acupressure points including 2 points in the upper/lower extremity along with the parallel points in each intervention.
  Arms: acupressure

SUMMARY:
The study was conducted randomly controlled to determine the effect of acupressure application on menopausal complaints among women who applied to Cancer Early Diagnosis and Screening Center.

DETAILED DESCRIPTION:
Research, between September 2019 and February 2020 of cancer in the body healthy life center in the east of the provincial center of Turkey was held by early diagnosis and screening center that refer to women.

The Universe and Sample of the Research The universe of the study consisted of women who applied to cancer early diagnosis and screening center for examination for any reason.

The calculation of the sample size of the study was determined according to the studies in which non-pharmacological methods were used to cope with menopausal symptoms. The calculation was determined according to the effect size of 0.5 in a moderate level, considering the effect size ranging between (0.25-0.83) reported by the studies on the subject.

ELIGIBILITY:
Inclusion Criteria:

* in the 45-65 age range.

Exclusion Criteria:

* receiving pharmacological treatment related to menopause,
* having a communication problem,
* have a hearing problem
* It is the presence of tissue deformity in its extremities.

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 120 (Actual)
Dates: Start 2019-06-05 (Actual); Primary Completion 2019-09-13 (Actual); Study Completion 2020-02-25 (Actual)

PRIMARY OUTCOMES:
Effect of Acupressure Application on Menopausal Symptoms | 8 week
  Menopause Rating Scale

CONTACTS AND LOCATIONS:
Locations (1):
- Didem Simsek Kucukkelepce, Adıyaman, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided